CLINICAL TRIAL: NCT01300234
Title: A Multi-centre, Double Blind, Double Dummy, Randomised, Controlled Study to Evaluate the Efficacy and Safety of TDF 300mg Once Daily (QD) Versus Adefovir Dipivoxil (ADV) 10mg QD in Chinese Subjects With CHB
Brief Title: Efficacy and Safety of Tenofovir Disoproxil Fumarate (TDF) 300mg in Chinese Subjects With Chronic Hepatitis B (CHB)
Acronym: TDF in CHB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114648
Record Dates: First submitted 2011-02-03; First posted 2011-02-21 (Estimated); Results first posted 2013-08-16 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis B
Keywords: tenofovir disoproxil fumarate; chronic hepatitis B; adefovir dipivoxil
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — Tenofovir; Tablets; adefovir dipivoxil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (TDF tablets) (Experimental): Tenofovir disoproxil fumarate (TDF) tablets
  Interventions: Drug: Tenofovir disoproxil fumarate (TDF) tablets
- B (ADV tablets) (Active Comparator): Adefovir dipivoxil (ADV) tablets
  Interventions: Drug: Adefovir dipivoxil (ADV) tablets

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate (TDF) tablets — white, almond-shaped, film-coated tablets containing 300mg of TDF
  Other Names: TDF tablet
  Arms: A (TDF tablets)
Drug: Adefovir dipivoxil (ADV) tablets — white to off-white, round, biconvex tablets containing 10mg of ADV
  Other Names: ADV tablet
  Arms: B (ADV tablets)

SUMMARY:
This is a multi-centre, double blind, double dummy, randomised, controlled study to evaluate the efficacy and safety of TDF 300mg QD versus ADV 10mg QD in Chinese subjects with CHB. This study is designed to demonstrate the superiority of TDF 300mg QD over ADV 10mg QD in treating Chinese subjects with CHB (hepatitis B e antigen [HBeAg] positive subjects and HBeAg negative subjects). It will also provide long-term efficacy and safety data (up to 240 weeks) for TDF 300 mg administered once daily.

DETAILED DESCRIPTION:
This is a multi-centre, double-blind, double-dummy, randomised, controlled study to evaluate the efficacy and safety of TDF 300mg QD versus ADV 10mg QD in Chinese subjects with CHB. Four hundred and ninety-four subjects with CHB (200 HBeAg positive subjects and 294 HBeAg negative subjects) will be randomised (1:1ratio) to either TDF 300mg QD or ADV 10mg QD treatment arms. The primary endpoint is the proportion of subjects with blood hepatitis B virus (HBV) deoxyribonucleic acid (DNA) <400copies/mL (Roche COBAS Taqman HBV test) at Week 48 in HBeAg positive subjects with CHB and HBeAg negative subjects with CHB. This is a two-part study. The first treatment period (baseline to Week 48) will investigate the effects of TDF and ADV on safety and efficacy endpoints; dosing will be double-blind. This period will be followed by 192 weeks in which all subjects will receive open-label TDF (Week 49 to Week 240). Subjects will undergo regular safety and efficacy assessments every 4 weeks for the first 12 weeks followed by every 12 weeks for a total of up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg positive/negative CHB with blood HBVDNA≥10^5 copies/mL and elevated ALT
* Nucleoside and nucleotide naïve CHB subjects. Previous lamivudine treatment is allowed in less than 10% of the total study population

Exclusion Criteria:

* subjects with hepatocellular carcinoma (HCC) potential or decompensated liver disease
* subjects with acute liver disease due to other causes
* subjects with medication history of immunosuppressive therapy, immunomodulatory therapy, systemic cytotoxic agents, chronic antiviral agents including Chinese herbal medicines known to have activity against HBV (e.g., lamivudine, hepatitis B immunoglobulin (HBIg)) within the previous 6 months prior to randomisation into this study

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2011-03-30 (Actual); Primary Completion 2012-10-17 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- China (12):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Shanghai

REFERENCES:
- [Derived] Liang X, Gao Z, Xie Q, Zhang J, Sheng J, Cheng J, Chen C, Mao Q, Zhao W, Ren H, Tan D, Niu J, Chen S, Pan C, Tang H, Wang H, Mao Y, Jia J, Ning Q, Xu M, Wu S, Li J, Zhang X, Zhang W, Xiong C, Hou J. Long-term efficacy and safety of tenofovir disoproxil fumarate in Chinese patients with chronic hepatitis B: 5-year results. Hepatol Int. 2019 May;13(3):260-269. doi: 10.1007/s12072-019-09943-6. Epub 2019 Apr 11. PMID 30977033
- [Derived] Hou JL, Gao ZL, Xie Q, Zhang JM, Sheng JF, Cheng J, Chen CW, Mao Q, Zhao W, Ren H, Tan DM, Niu JQ, Chen SJ, Pan C, Tang H, Wang H, Mao YM, Jia JD, Ning Q, Xu M, Wu SM, Li J, Zhang XX, Ji Y, Dong J, Li J. Tenofovir disoproxil fumarate vs adefovir dipivoxil in Chinese patients with chronic hepatitis B after 48 weeks: a randomized controlled trial. J Viral Hepat. 2015 Feb;22(2):85-93. doi: 10.1111/jvh.12313. Epub 2014 Sep 22. PMID 25243325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2 sequential treatment period study. In first period (double-blinded),participants received tenofovir disoproxil fumarate (TDF) 300 milligram (mg) once daily (QD) or adefovir dipivoxil (ADV) 10 mg QD for 48 Weeks. In second period (open-label single treatment), participants received TDF 300 mg QD for additional 192 Weeks.
Pre-assignment Details: 969 participants were screened, 512 were randomized and 509 were treated with at least one dose of study medication in the double-blind treatment period. Participants who received at least one dose of study medication continued in open-label period.
Groups:
- TDF-TDF: In first double-blinded treatment period, participants self-administered TDF 300 mg tablets plus matching ADV placebo at the same time QD for 48 Weeks. In second open-label treatment period, participants self-administered TDF 300 mg QD for additional 192 Weeks.
- ADV-TDF: In first double-blinded treatment period, participants self-administered ADV 10 mg tablets plus matching TDF placebo at the same time QD for 48 Weeks. In second open-label treatment, participants self-administered TDF 300 mg QD for additional 192 Weeks.
Period: Overall Study
Arm/Group | TDF-TDF | ADV-TDF
Started | 257 | 255
Completed | 229 | 228
Not Completed | 28 | 27
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Lost to Follow-up | 14 | 12
Not completed — Pregnancy | 2 | 1
Not completed — Participant reached stopping critera | 2 | 0
Not completed — Participant stopped medication | 1 | 1
Not completed — Participant refused return to hospital | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were collected in members of the Intent-to-Treat Population, comprised of all randomized participants who received at least one dose of study medication.
Groups:
- TDF-TDF: In first treatment period, participants self-administered TDF 300 mg tablets plus matching ADV placebo at the same time QD for 48 Weeks. In second treatment, participants self-administered TDF 300 mg QD for additional 192 Weeks.
- ADV-TDF: In first treatment period, participants self-administered ADV 10 mg tablets plus matching TDF placebo at the same time QD for 48 Weeks. In second treatment, participants self-administered TDF 300 mg QD for additional 192 Weeks.
- Total: Total of all reporting groups
Arm/Group | TDF-TDF | ADV-TDF | Total
Number analyzed (Participants) | 257 | 252 | 509
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all randomized participants who received at least one dose of study medication.
  Years | 36.1 (10.48) | 36.4 (10.43) | 36.3 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all randomized participants who received at least one dose of study medication.
  Participants
    Female | 43 | 42 | 85
    Male | 214 | 210 | 424
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all randomized participants who received at least one dose of study medication.
  participants
    Asian - East Asian Heritage | 257 | 252 | 509

OUTCOME MEASURES:

1. Primary Outcome: Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) <400 Copies/Milliliter (mL) at Week 48
Description: The number of participants with Hepatitis B Virus (HBV) deoxyribonucleic acid (DNA) <400 copies/milliliter (mL) at Week 48 in the hepatitis B e antigen (HBeAg)-positive and HBeAg-negative population was assessed. HBeAg is a viral protein that is secreted by hepatitis B-infected cells. It is associated with chronic hepatitis B infections and is used as a marker of active viral disease and a participant's degree of infectiousness. A positive result indicates that the participant has high levels of virus in the blood and greater infectiousness. Usually, a negative result indicates that the participant has lower levels of virus in the blood and is less infectious. A "non-completers equal failures" approach is used for the analysis in ITT population. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Week 48
Population: Intent-to-Treat (ITT) Population: All randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Groups:
- TDF 300 mg: Participants self-administered TDF 300 mg tablets plus matching ADV placebo at the same time QD for 48 Weeks.
- ADV 10 mg: Participants self-administered ADV 10 mg tablets plus matching TDF placebo at the same time QD for 48 Weeks.
Arm/Group | TDF 300 mg | ADV 10 mg
Number analyzed (Participants) | 257 | 252
Participants
  HBeAg-positive, n=103, 99: number analyzed (Participants) | 103 | 99
  HBeAg-positive, n=103, 99 | 79 | 18
  HBeAg-negative, n=154, 153: number analyzed (Participants) | 154 | 153
  HBeAg-negative, n=154, 153 | 149 | 109
Statistical Analysis 1: Comparison: TDF 300 mg vs ADV 10 mg; Test type: Superiority or Other; p < 0.0001, Roche COBAS Taqman HBV test — HBeAg-positive participants; percentage of participants = 58.5, 97.5% CI 2-sided [45.8 to 71.3] — A "non-completers equal failures" approach is used for the primary analysis. The estimated value represents the difference between the percentage of participants achieving HBV DNA <400 copies/mL at Week 48 in the TDF group and the ADV group
Statistical Analysis 2: Comparison: TDF 300 mg vs ADV 10 mg; Test type: Superiority or Other; p < 0.0001, Roche COBAS Taqman HBV test — HBeAg-negative participants; percentage of participants = 25.6, 97.5% CI 2-sided [16.7 to 34.3] — A "non-completers equal failures" approach was used for the primary analysis. The estimated value represents the difference between the percentage of participants achieving HBV DNA <400 copies/mL at Week 48 in the TDF group and the ADV group

2. Secondary Outcome: Participants With HBV DNA <400 Copies/mL at Weeks 96, 144, 192, and 240
Description: The number of participants with HBV DNA <400 copies/mL in the hepatitis B e antigen (HBeAg)-positive and HBeAg-negative population was assessed. HBeAg is a viral protein that is secreted by hepatitis B-infected cells. It is associated with chronic hepatitis B infections and is used as a marker of active viral disease and a participant's degree of infectiousness. A positive result indicates that the participant has high levels of virus in the blood and greater infectiousness. Usually, a negative result indicates that the participant has lower levels of virus in the blood and is less infectious. Week 96, 144, 192, and 240 data are not yet available, as this report includes data up to and including Week 48. A "non-completers equal failures" approach is used for the analysis in ITT population. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Weeks 96, 144, 192, and 240
Population: ITT Population
Measure: Number; unit: Participants
Groups:
- ADV-TDF: In first double-blinded treatment period, participants self-administered ADV 10 mg tablets plus matching TDF placebo at the same time QD for 48 Weeks. In second open-label treatment period, participants self-administered TDF 300 mg QD for additional 192 Weeks.
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
Participants
  Week 96, HBeAg-positive, n=103, 99: number analyzed (Participants) | 103 | 99
  Week 96, HBeAg-positive, n=103, 99 | 95 | 92
  Week 96, HBeAg-negative, n=154, 153: number analyzed (Participants) | 154 | 153
  Week 96, HBeAg-negative, n=154, 153 | 144 | 143
  Week 144, HBeAg-positive, n=103, 99: number analyzed (Participants) | 103 | 99
  Week 144, HBeAg-positive, n=103, 99 | 97 | 95
  Week 144, HBeAg-negative, n=154,153: number analyzed (Participants) | 154 | 153
  Week 144, HBeAg-negative, n=154,153 | 144 | 145
  Week 192, HBeAg-positive, n=103,99: number analyzed (Participants) | 103 | 99
  Week 192, HBeAg-positive, n=103,99 | 94 | 93
  Week 192,HBeAg-negative, n=154,153: number analyzed (Participants) | 154 | 153
  Week 192,HBeAg-negative, n=154,153 | 144 | 141
  Week 240, HBeAg-positive, n=103,99: number analyzed (Participants) | 103 | 99
  Week 240, HBeAg-positive, n=103,99 | 87 | 87
  Week 240, HBeAg-negative, n=154,153: number analyzed (Participants) | 154 | 153
  Week 240, HBeAg-negative, n=154,153 | 138 | 137

3. Secondary Outcome: Change From Baseline of Log 10 Copies/mL HBV DNA at Weeks 48, 96, 144, 192 and 240
Description: Change from Baseline of log 10 copies/mL HBV DNA at Weeks 48, 96, 144, 192 and 240 in the HBeAg-positive and HBeAg-negative population was assessed. HBeAg is a viral protein that is secreted by hepatitis B-infected cells. It is associated with chronic hepatitis B infections and is used as a marker of active viral disease and a participant's degree of infectiousness. A positive result indicates that the participant has high levels of virus in the blood and greater infectiousness. Usually a negative result indicates that the participant has lower levels of virus in the blood and less infectious. Values at Day 0 were considered as Baseline values. Change from Baseline was calculated as post Baseline values minus Baseline values. A "non-completers equal failures" approach is used for the analysis in ITT population. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline, Weeks 48, 96, 144, 192 and 240
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
log10 copies/mL
  Week 48,HBeAg-positive, n=102, 97: number analyzed (Participants) | 102 | 97
  Week 48,HBeAg-positive, n=102, 97 | -6.4 (0.86) | -4.4 (1.69)
  Week 48,HBeAg-negative, n=151, 148: number analyzed (Participants) | 151 | 148
  Week 48,HBeAg-negative, n=151, 148 | -4.9 (1.16) | -4.3 (1.31)
  Week 96, HBeAg-positive, n=101, 97: number analyzed (Participants) | 101 | 97
  Week 96, HBeAg-positive, n=101, 97 | -6.5 (0.86) | -6.5 (0.81)
  Week 96, HBeAg-negative, n=147,148: number analyzed (Participants) | 147 | 148
  Week 96, HBeAg-negative, n=147,148 | -4.9 (1.26) | -4.8 (1.17)
  Week 144, HBeAg-postive, n=100, 96: number analyzed (Participants) | 100 | 96
  Week 144, HBeAg-postive, n=100, 96 | -6.6 (0.86) | -6.5 (0.80)
  Week 144, HBeAg-negative, n=145, 146: number analyzed (Participants) | 145 | 146
  Week 144, HBeAg-negative, n=145, 146 | -4.9 (1.16) | -4.9 (1.09)
  Week 192, HBeAg-positive, n=97,93: number analyzed (Participants) | 97 | 93
  Week 192, HBeAg-positive, n=97,93 | -6.6 (0.86) | -6.6 (0.81)
  Week 192, HBeAg-negative, n=145,145: number analyzed (Participants) | 145 | 145
  Week 192, HBeAg-negative, n=145,145 | -4.9 (1.17) | -4.8 (1.14)
  Week 240, HBeAg-positive, n=91,90: number analyzed (Participants) | 91 | 90
  Week 240, HBeAg-positive, n=91,90 | -6.6 (1.01) | -6.5 (0.79)
  Week 240, HBeAg-negative, n=138,138: number analyzed (Participants) | 138 | 138
  Week 240, HBeAg-negative, n=138,138 | -4.9 (1.16) | -4.9 (1.07)

4. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normalization at Weeks 48, 96, 144, 192 and 240 in Participants Who Had Abnormal ALT at Baseline
Description: Participants who had abnormal ALT at Baseline and had normalized ALT at Weeks 48, 96, 144, 192 and 240 were assessed. This report includes data up to and including Weeks 48, 96, 144, 192 and 240. An increased level of ALT is referred to as abnormal ALT (the normal range is 0 to 48 units per liter [U/L]). Values at Day 0 were considered as Baseline values. A "non-completers equal failures" approach is used for the analysis in ITT population. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline; Weeks 48, 96, 144, 192 and 240
Population: ITT Population.
Measure: Number; unit: Participants
Groups:
- TDF-TDF: In first double-blinded treatment period, participants self-administered TDF 300 mg tablets plus matching ADV placebo at the same time QD for 48 Weeks. In second open-label treatment period, participants self-administered TDF 300 mg once daily for additional 192 Weeks.
- ADV-TDF: In first double-blinded treatment period, participants self-administered ADV 10 mg tablets plus matching TDF placebo at the same time QD for 48 Weeks. In second open-label treatment period, participants self-administered TDF 300 mg once daily for additional 192 Weeks.
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
Participants
  Week 48, HBeAg-positive, n=102, 97: number analyzed (Participants) | 102 | 97
  Week 48, HBeAg-positive, n=102, 97 | 88 | 83
  Week 48, HBeAg-negative, n=136, 132: number analyzed (Participants) | 136 | 132
  Week 48, HBeAg-negative, n=136, 132 | 120 | 116
  Week 96, HBeAg-positive, n=102, 97: number analyzed (Participants) | 102 | 97
  Week 96, HBeAg-positive, n=102, 97 | 93 | 88
  Week 96, HBeAg-negative, n=136,132: number analyzed (Participants) | 136 | 132
  Week 96, HBeAg-negative, n=136,132 | 126 | 118
  Week 144, HBeAg-positive, n=102, 97: number analyzed (Participants) | 102 | 97
  Week 144, HBeAg-positive, n=102, 97 | 92 | 87
  Week 144, HBeAg-negative, n=136, 132: number analyzed (Participants) | 136 | 132
  Week 144, HBeAg-negative, n=136, 132 | 123 | 119
  Week 192, HBeAg-positive, n=102, 97: number analyzed (Participants) | 102 | 97
  Week 192, HBeAg-positive, n=102, 97 | 89 | 79
  Week 192, HBeAg-negative, n=136,132: number analyzed (Participants) | 136 | 132
  Week 192, HBeAg-negative, n=136,132 | 125 | 118
  Week 240, HBeAg-positive, n=102, 97: number analyzed (Participants) | 102 | 97
  Week 240, HBeAg-positive, n=102, 97 | 82 | 80
  Week 240, HBeAg-negative, n=136,132: number analyzed (Participants) | 136 | 132
  Week 240, HBeAg-negative, n=136,132 | 119 | 111

5. Secondary Outcome: Number of Participants With Histological Improvement at Weeks 48 and 240 Who Had a Baseline Knodell Necroinflammatory Score (KNS) >=2.
Description: Histological improvement is defined as a reduction of >=2 points in the KNS with no increase in fibrosis at Week 48 and Week 240 in participants with Baseline KNS >=2 which was derived from the American Association for the Study of Liver Diseases Practice Guidelines for Management of Chronic Hepatitis B (2009) and the European Association for the Study of the Liver Clinical Practice Guidelines Management of chronic hepatitis B virus infection (2012). The Knodell scale consists of 5 domains: periportal +/- bridging necrosis (scored from best to worst: 0, 1, 3, 4, 5, 6, or 10); intralobular degeneration and focal necrosis (0 to 4); portal inflammation (0 to 4); and fibrosis (0 to 4). The necroinflammatory score (ranging from 0 [best] to 14 [worst]) is the combined score for necrosis (0 to 10) plus inflammation (0 to 4; the participant is scored for only one inflammatory condition). Liver biopsy slides within 6 months prior to randomization could be accepted as Baseline evaluation.
Time Frame: Baseline; Week 48 and Week 240
Population: ITT Population. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Measure: Number; unit: Participants
Groups:
- TDF-TDF: In first treatment double-blinded period, participants self-administered TDF 300 mg tablets plus matching ADV placebo at the same time QD for 48 Weeks. In second open-label treatment period, participants self-administered TDF 300 mg QD for additional 192 Weeks.
- ADV-TDF: In first treatment double-blinded period, participants self-administered ADV 10 mg tablets plus matching TDF placebo at the same time QD for 48 Weeks. In second open-label treatment period, participants self-administered TDF 300 mg QD for additional 192 Weeks.
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 86 | 102
Participants
  Week 48, HBeAg-positive, n=38, 49: number analyzed (Participants) | 38 | 49
  Week 48, HBeAg-positive, n=38, 49 | 31 | 39
  Week 48, HBeAg-negative, n=45, 50: number analyzed (Participants) | 45 | 50
  Week 48, HBeAg-negative, n=45, 50 | 32 | 34
  Week 240, HBeAg-positive, n=38, 49: number analyzed (Participants) | 38 | 49
  Week 240, HBeAg-positive, n=38, 49 | 5 | 2
  Week 240, HBeAg-negative, n=45, 50: number analyzed (Participants) | 45 | 50
  Week 240, HBeAg-negative, n=45, 50 | 8 | 4

6. Secondary Outcome: Number of HBeAg-positive Participants Achieving HBeAg Loss and HBeAg Seroconversion at Weeks 24, 48, 96, 144, 192 and 240.
Description: HBeAg loss is defined as a negative HBeAg result for those participants who were HBeAg positive at Baseline. Seroconversion to anti-HBe is defined as HBeAg loss and a positive anti-HBe result. This report includes data up to and including Weeks 24, 48, 96, 144, 192 and 240.
Time Frame: Weeks 24, 48, 96, 144, 192 and 240
Population: ITT Population. Only those participants with data available at specific time point were analyzed
Measure: Number; unit: Participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 103 | 99
Participants
  Week 24, HBeAg loss | 15 | 4
  Week 24, HBeAg seroconversion | 14 | 4
  Week 48, HBeAg loss | 18 | 10
  Week 48, HBeAg seroconversion | 16 | 9
  Week 96, HBeAg loss | 37 | 21
  Week 96, HBeAg seroconversion | 32 | 18
  Week 144, HBeAg loss | 37 | 24
  Week 144, HBeAg seroconversion | 33 | 20
  Week 192, HBeAg loss | 43 | 31
  Week 192, HBeAg seroconversion | 33 | 24
  Week 240, HBeAg loss | 43 | 36
  Week 240, HBeAg seroconversion | 33 | 28

7. Secondary Outcome: Number of HBeAg-positive Participants Achieving Hepatitis B Surface Antigen (HBsAg) Loss and HBsAg Seroconversion at Weeks 24, 48, 96, 144, 192 and 240
Description: HBsAg loss is defined as negative HBsAg results for those participants with who were HBsAg positive at Baseline. Seroconversion to anti-HBs is defined as HBsAg loss and a positive anti-HBs result. This report includes data up to and including Week 240.
Time Frame: Weeks 24, 48, 96, 144, 192 and 240
Population: ITT Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 103 | 99
Participants
  Week 24, HBsAg loss | 0 | 0
  Week 24, HBsAg seroconversion | 0 | 0
  Week 48, HBsAg loss | 0 | 0
  Week 48, HBsAg seroconversion | 0 | 0
  Week 96, HBsAg loss | 0 | 0
  Week 96, HBsAg seroconversion | 0 | 0
  Week 144, HBsAg loss | 1 | 0
  Week 144, HBaAg seroconversion | 0 | 0
  Week 192, HBsAg, loss | 1 | 0
  Week 192, HBsAg, seroconversion | 0 | 0
  Week 240, HBsAg loss | 1 | 0
  Week 240 HBsAg seroconversion | 0 | 0

8. Secondary Outcome: Number of HBeAg-negative Participants Achieving HBsAg Loss and HBsAg Seroconversion at Weeks 24, 48, 96, 144, 192, 240
Description: HBsAg loss is defined as a negative HBsAg result for those participants with who were HBsAg positive at Baseline. Seroconversion to anti-HBs is defined as HBsAg loss and a positive anti-HBs result. This report includes data up to and including Week 240.
Time Frame: Weeks 24, 48, 96, 144, 192 and 240
Population: ITT Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 154 | 153
Participants
  Week 24, HBsAg loss | 0 | 0
  Week 24, HBsAg seroconversion | 0 | 0
  Week 48, HBsAg loss | 0 | 0
  Week 48, HBsAg seroconversion | 0 | 0
  Week 96, HBsAg loss | 0 | 0
  Week 96, HBsAg seroconversion | 0 | 0
  Week 144, HBsAg loss | 0 | 1
  Week 144, HBsAg seroconversion | 0 | 1
  Week 192, HBsAg loss | 0 | 0
  Week 192, HBsAg seroconversion | 0 | 0
  Week 240, HBsAg loss | 0 | 0
  Week 240, HBsAg seroconversion | 0 | 0

9. Secondary Outcome: Number of Participants Achieving Durable HBsAg Loss From Weeks 24 to Week 48
Description: Durable HBsAg loss is defined as the loss of HBsAg and no detectable HBV DNA and ALT normalization at any three consecutive visits at least 12 Weeks apart. This report includes data up to and including Week 48. A "non-completers equal failures" approach was used for the analysis in ITT population.
Time Frame: Week 24 to Week 48
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg | ADV 10 mg
Number analyzed (Participants) | 257 | 252
Participants
  HBeAg-positive, n =100, 97: number analyzed (Participants) | 100 | 97
  HBeAg-positive, n =100, 97 | 0 | 0
  HBeAg-negative, n=150, 147: number analyzed (Participants) | 150 | 147
  HBeAg-negative, n=150, 147 | 0 | 0

10. Secondary Outcome: Number of Participants Achieving Durable HBsAg Loss From Weeks 96 to Week 240
Description: Durable HBsAg loss is defined as the loss of HBsAg and no detectable HBV DNA and ALT normalization at any three consecutive visits at least 12 Weeks apart from Week 96 to 240. This report includes data up to and including Week 240. A "non-completers equal failures" approach was used for the analysis in ITT population.
Time Frame: Week 96 to Week 240
Population: ITT Population.
Measure: Number; unit: Participants
Groups:
- ADV-TDF: In first double-blinded treatment, participants self-administered ADV 10 mg tablets plus matching TDF placebo at the same time QD for 48 Weeks. In second open-label treatment period, participants self-administered TDF 300 mg QD for additional 192 Weeks.
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
Participants
  HBeAg-positive, n= 88, 90: number analyzed (Participants) | 88 | 90
  HBeAg-positive, n= 88, 90 | 1 | 0
  HBeAg-negative, n = 132, 137: number analyzed (Participants) | 132 | 137
  HBeAg-negative, n = 132, 137 | 0 | 1

11. Secondary Outcome: Number of Participants With Virological Breakthrough at Weeks 48, 96, 144, 192 and 240
Description: The number of HBeAg-positive and HBeAg-negative participants who had virological breakthrough at Weeks 48, 96, 144, 192 and 240 were assessed. Virological breakthrough is defined by >= one log increase in HBV DNA from NADIR (as determined by two sequential HBV DNA measurements at least one month apart or last on treatment measurement). A "non-completers equal failures" approach was used for the analysis in ITT population.
Time Frame: Weeks 48, 96, 144, 192 and 240
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
Participants
  Week 48,HBeAg-Positive, n=103, 99: number analyzed (Participants) | 103 | 99
  Week 48,HBeAg-Positive, n=103, 99 | 0 | 4
  Week 48, HBeAg-Negative, n=154, 153: number analyzed (Participants) | 154 | 153
  Week 48, HBeAg-Negative, n=154, 153 | 0 | 2
  Week 96, HBeAg-positive, n=103, 99: number analyzed (Participants) | 103 | 99
  Week 96, HBeAg-positive, n=103, 99 | 0 | 4
  Week 96, HBeAg-negative, n=154, 153: number analyzed (Participants) | 154 | 153
  Week 96, HBeAg-negative, n=154, 153 | 2 | 3
  Week 144, HBeAg-positive, n=103, 99: number analyzed (Participants) | 103 | 99
  Week 144, HBeAg-positive, n=103, 99 | 0 | 7
  Week 144, HBeAg-negative, n=154, 153: number analyzed (Participants) | 154 | 153
  Week 144, HBeAg-negative, n=154, 153 | 3 | 4
  Week 192, HBeAg-positive, n=103, 99: number analyzed (Participants) | 103 | 99
  Week 192, HBeAg-positive, n=103, 99 | 0 | 7
  Week 192, HBeAg-negative, n=154, 153: number analyzed (Participants) | 154 | 153
  Week 192, HBeAg-negative, n=154, 153 | 3 | 5
  Week 240, HBeAg-positive, n=103, 99: number analyzed (Participants) | 103 | 99
  Week 240, HBeAg-positive, n=103, 99 | 4 | 11
  Week 240, HBeAg-negative, n=154, 153: number analyzed (Participants) | 154 | 153
  Week 240, HBeAg-negative, n=154, 153 | 3 | 8

12. Secondary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Any Non-serious Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is Grade 4 (life threatening or disabling). Participants with any non-serious AEs and SAEs has been reported.
Time Frame: Up to Week 240 treatment period and 24 weeks follow-up visit off treatment
Population: Safety Analysis Population: All participants who received at least one dose of study medication and had at least one post-Baseline safety assessment
Measure: Number; unit: Participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
Participants
  Non-serious AE | 140 | 121
  SAE | 12 | 20

13. Secondary Outcome: Number of Participants With the Indicated Grade 3 and Grade 4 Treatment-emergent (TE) Laboratory Abnormalities (LAs)
Description: TE grade 3 or grade 4 LAs are defined as values that increase by >=1 grade from Baseline (Day 0) to Grade 3 (severe) or 4 (potentially life threatening) at any post-Baseline value. The Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities, version 21, September 2011 was referred for grading. Laboratory parameters assessed included Sodium for hyponatremia and hypernatremia; Potassium for hypokalemia and hyperkalemia; glucose for hypoglycemia and hyperglycemia non-fasting; Phosphate for hypophosphatemia; alanine aminotransferase/aspartate aminotransferase, bilirubin, creatinine kinase, hemoglobin, platelets, neutrophils, lymphocytes, prothrombin time and amylase.
Time Frame: Up to Week 240
Population: Safety Analysis Population
Measure: Number; unit: participants
Groups:
- TDF-TDF: In first double-blinded treatment period, participants self-administered TDF 300 mg tablets plus matching ADV placebo at the same time QD for 48 Weeks.In second open-label treatment period, participants self-administered TDF 300 mg QD for additional 192 Weeks.
- ADV-TDF: In first double-blinded treatment period, participants self-administered ADV 10 mg tablets plus matching TDF placebo at the same time QD for 48 Weeks.In second open-label treatment period, participants self-administered TDF 300 mg QD for additional 192 Weeks.
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
participants
  Sodium | 2 | 0
  Phosphate | 2 | 3
  Alanine aminotransferase | 19 | 14
  Aspartate aminotransferase | 10 | 6
  Bilirubin | 1 | 1
  Creatine kinase | 6 | 4
  Hemoglobin | 4 | 5
  Platelets | 4 | 3
  Neutrophils | 6 | 4
  Prothrombin time | 10 | 17
  Potassium | 1 | 0
  Glucose | 1 | 2
  Lymphocytes | 2 | 3
  Amylase | 1 | 2

14. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Laboratory Abnormalities for Serum Creatinine and Serum Phosphorus
Description: The Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities, version 21, September 2011 was referred for grading. Serum creatinine: Grade 1, > 133 to 177 micromoles per Liter (µmoles/Liter), Grade 2, >177 to 265 µmoles/Liter, Grade 3, >265 to 530 µmoles/Liter, Grade 4, >530 µmoles/Liter. Serum phosphorus: Grade 2, 0.63 to <0.80 millimoles per Liter (mmoles/L), Grade 3, 0.31 to <0.63 mmoles/L, Grade 4, <0.31 mmoles/L. The normal range for serum phosphorus was 0.8 to 1.45 mmoles/L; the upper limit for a Grade 2 abnormality is 0.80 mmoles/L. Therefore, no Grade 1 abnormalities could be attributed, as values were contained within the normal range. NA indicates the value was not available for the indicated time point.
Time Frame: Up to Week 240
Population: Safety Analysis Population
Measure: Number; unit: Participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
Participants
  Serum creatinine, Grade 1 | 0 | 1
  Serum creatinine, Grade 2 | 0 | 0
  Serum creatinine, Grade 3 | 0 | 0
  Serum creatinine, Grade 4 | 0 | 0
  Serum phosphorus, Grade 1 | NA — The normal range for serum phosphorus was 0.8-1.45 mmol/L; the upper limit for a Grade 2 abnormality was 0.80 mmol/L. Therefore, no Grade 1 abnormalities could be attributed as values were contained within the normal range. | NA — The normal range for serum phosphorus was 0.8-1.45 mmol/L; the upper limit for a Grade 2 abnormality was 0.80 mmol/L. Therefore, no Grade 1 abnormalities could be attributed as values were contained within the normal range.
  Serum phosphorus, Grade 2 | 42 | 55
  Serum phosphorus, Grade 3 | 2 | 3
  Serum phosphorus, Grade 4 | 0 | 0

15. Secondary Outcome: Number of Participants in the Indicated Category for Renal Laboratory Abnormalities
Description: The Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities, version 21, September 2011 was used for grading. "Confirmed" is defined as two consecutive visits. mg=milligrams. dL=deciliter, G= Grade.
Time Frame: Up to Week 240
Population: Safety Analysis Population
Measure: Number; unit: Participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 257 | 252
Participants
  Creatinine increase of 0.5 mg/dL above Baseline | 1 | 0
  Confirmed creatinine >=2.0 mg/dL | 0 | 0
  Confirmed clearance <50 milliliters/minute | 0 | 0
  Confirmed phosphorus G 3/4 abnormality, <2.0 mg/dL | 3 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment up to 240 weeks treatment period and 24 weeks follow-up visit off treatment.
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the Safety Analysis (SA) Population, comprised of all participants who received at least one dose of study medication and had at least one post-Baseline safety assessment.
Arm/Group | TDF-TDF | ADV-TDF
All-Cause Mortality (participants affected / at risk) | 1/257 | 0/252
Serious Adverse Events (participants affected / at risk) | 12/257 | 20/252
Other Adverse Events (participants affected / at risk) | 140/257 | 121/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDF-TDF (N=257) | ADV-TDF (N=252)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Miscarriage of partner (Social circumstances) | 0 | 1
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDF-TDF (N=257) | ADV-TDF (N=252)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5
Alanine aminotransferase increased (Investigations) | 16 | 8
Asthenia (General disorders) | 4 | 5
Bronchitis (Infections and infestations) | 1 | 4
Cholelithiasis (Hepatobiliary disorders) | 5 | 4
Dizziness (Nervous system disorders) | 2 | 4
Gallbladder polyp (Hepatobiliary disorders) | 6 | 4
Gingivitis (Infections and infestations) | 3 | 2
Hepatic pain (Hepatobiliary disorders) | 5 | 5
Hepatic steatosis (Hepatobiliary disorders) | 11 | 11
Nasopharyngitis (Infections and infestations) | 8 | 8
Nephrolithiasis (Renal and urinary disorders) | 5 | 13
Upper respiratory tract infection (Infections and infestations) | 34 | 25
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Accessory spleen (Congenital, familial and genetic disorders) | 0 | 1
Hamartoma (Congenital, familial and genetic disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1
Hypogonadism (Endocrine disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 2
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 1
Chest discomfort (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 3
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 1
Sensation of foreign body (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 3 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 2
Hepatitis (Hepatobiliary disorders) | 2 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1
Perihepatic discomfort (Hepatobiliary disorders) | 1 | 4
Food allergy (Immune system disorders) | 1 | 0
Eczema infected (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 3 | 4
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 2
Tonsillitis (Infections and infestations) | 2 | 0
Tonsillitis bacterial (Infections and infestations) | 0 | 1
Viral rash (Infections and infestations) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Alpha 1 foetoprotein increased (Investigations) | 1 | 0
Amylase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 3
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine phosphokinase (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 7 | 8
Blood glucose increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 4 | 5
Blood potassium decreased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Hepatitis B DNA increased (Investigations) | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 1
Monocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 3 | 2
Prothrombin time prolonged (Investigations) | 3 | 2
Red blood cell count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Haemangioma of spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Headache (Nervous system disorders) | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0
Vascular headache (Nervous system disorders) | 0 | 1
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 4
Sleep disorder (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Nephrocalcinosis (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 6 | 3
Renal failure (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 2
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.